CLINICAL TRIAL: NCT03985826
Title: Health Care Utilisation Following Childhood Acute Lymphoblastic Leukaemia: A Matched Cohort Study
Brief Title: Health Care Utilisation Among Survivors of Childhood Acute Lymphoblastic Leukaemia
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other)
Responsible Party: Sponsor
Other Study IDs: ID277
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2019-06

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Childhood ALL survivors: The cohort of childhood ALL survivors will be identified in the Danish part of the Nordic Society of Paediatric Haematology and Oncology (NOPHO) ALL-Register .
  Interventions: Other: Diagnosis of and treatment for Acute lymphoblastic leukaemia in childhood
- Comparison cohort: A reference cohort (comparison cohort) of individuals will be sampled randomly from the source population matched by age and sex and without a history of childhood cancer in the calendar year where the case was diagnosed (density sampling). For each childhood ALL-patient we will choose ten comparison subjects.

INTERVENTIONS:
Other: Diagnosis of and treatment for Acute lymphoblastic leukaemia in childhood — The cohort of ALL survivors has all been diagnosed and treated for ALL in childhood
  Groups: Childhood ALL survivors

SUMMARY:
Improved understanding of the long-time healthcare utilisation of childhood cancer survivors is relevant as it can be seen as a proxy for the population's morbidity.

The investigators will conduct a historic population-based matched cohort study using Danish nationwide registry data. Eligible children are children 1.0-17.9 years diagnosed with Acute lymphoblastic leukaemia (ALL) in Denmark from 1994 till 2016. The primary outcome is yearly contact rates to primary healthcare.

DETAILED DESCRIPTION:
Acute lymphoblastic leukaemia (ALL) is the most frequent single form of cancer in children accounting for 40-45 new cases every year in Denmark. Over the past decades, advances in treatment have led to an increasing number of children who survive cancer and more than 80% of children with ALL now become long-term survivors. This means a growing population of childhood ALL survivors. In survivors, the cancer itself and treatment late-effects can lead to ongoing health care use.

Register studies of long-term survivors of childhood cancer have shown an increased risk of hospitalisation compared to the general population. It is mentioned in many of the studies that contact rates could be underestimated when looking at hospital contacts only.

The literature about non-hospital-based contacts with a doctor in childhood cancer survivors is scarce.

ELIGIBILITY:
Inclusion Criteria:

* B-precursor ALL and T-ALL enrolled in the NOPHO ALL-92, ALL-2000 and ALL-2008 trials.
* Treated at one of the four Danish paediatric oncology departments
* Age group 1.0-14.9 for the NOPHO ALL-92 and ALL-2000 trials. Age group 1.0-17.9 for the NOPHO ALL-2008 trial.
* Completed maintenance therapy in the time period form 01.01.1997 till 31.12.2016

Exclusion Criteria:

* Children with Down syndrome

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study population will be identified in the Danish part of the Nordic Society of Paediatric Haematology and Oncology ALL database.
  A reference cohort (comparison cohort) of individuals will be sampled randomly from the source population matched by age and sex and without a history of childhood cancer in the calendar year where the case was diagnosed (density sampling). For each childhood ALL-patient we will choose ten comparison subjects.
Sampling Method: Non-Probability Sample
Enrollment: 7348 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
The yearly contact rate to general practice for ALL survivors and controls | 1-20 years follow-up
  Analysing longitudinal health care data with analysis of both first and recurrent events

OTHER OUTCOMES:
The yearly contact rate to secondary healthcare for ALL survivors and controls | 1-20 years follow-up
  Analysing longitudinal health care data with analysis of both first and recurrent events

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vedsted, Professor, Study Director — Research Unit for General Practice, Institute for Public Health
Locations (1):
- Department of Public Health, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen KS, Klug Albertsen B, Schroder H, Zalounina Falborg A, Schmiegelow K, Rosthoj S, Callesen MT, Vedsted P. Health care utilisation following childhood acute lymphoblastic leukaemia: a population-based matched cohort study. BMJ Open. 2021 Nov 22;11(11):e049847. doi: 10.1136/bmjopen-2021-049847. PMID 34810184